CLINICAL TRIAL: NCT03980834
Title: Teachers Thriving Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-00204
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Social Emotional Competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Professional Learning, Program Training and Coaching (Active Comparator)
  Interventions: Behavioral: ParentCorps FUNdamentals; Behavioral: ParentCorps 101 E-learning; Behavioral: Training; Behavioral: Coaching
- Program for Parents of Pre-K Students (Active Comparator)
  Interventions: Behavioral: Training
- Program for Pre-K Students (Active Comparator)
  Interventions: Behavioral: Coaching

INTERVENTIONS:
Behavioral: ParentCorps FUNdamentals — is a series of large-group experiential PD days (in groups of 25-40 participants from across all schools) which takes place in the first summer prior to implementation. Leaders participate in a 2-day FUNdamentals series with leaders from other schools.
  Arms: Professional Learning, Program Training and Coaching
Behavioral: ParentCorps 101 E-learning — is a self-paced interactive web-based series with 7 modules intended to help facilitators build confidence and mastery of evidence-based practices.
  Arms: Professional Learning, Program Training and Coaching
Behavioral: Training — group-based series to prepare facilitators (mental health professionals and teachers) to implement Programs with fidelity and to ensure high levels of exposure by parents and students. Mental health professionals are supported to facilitate the Program for Parents (day and after-school versions) with fidelity. Pre-K teachers and assistants are supported to implement the Program for Students in the classroom. In addition, early childhood staff (including Kindergarten teachers as needed) is trained to facilitate the Program for Students during after-school hours in parallel with the Parenting Program. All facilitators receive training on engaging parents to participate
  Arms: Professional Learning, Program Training and Coaching; Program for Parents of Pre-K Students
Behavioral: Coaching — is one-on-one support provided in-vivo and from a distance (phone, text, email) to help users apply evidence-based practices in daily interactions with students and parents, and to support high levels of implementation fidelity and exposure. All Pre-K teachers and mental health professionals facilitating ParentCorps receive four on-site coaching visits and 10 30-minute calls for the remaining sessions in the first year for each cycle of implementation.
  Arms: Professional Learning, Program Training and Coaching; Program for Pre-K Students

SUMMARY:
This is a randomized, controlled, hybrid implementation-effectiveness design.whose primary aim is to examine the impact of ParentCorps plus Thrive Professional Learning, relative to Thrive Professional Learning and Inspire Professional Learning alone, on teachers' classroom teaching (knowledge, beliefs, skills and practice related to family engagement and social emotional learning) and teachers' social emotional development. The study also aims to understand the impact of Thrive Professional Learning versus Inspire Professional Learning alone on teachers and classrooms.

ELIGIBILITY:
Inclusion Criteria:

* The participants are lead teachers, assistant teachers, teaching assistants, paraprofessionals and teacher aides in 238 sites with Pre-K in NYC (for the purposes of this study, the term "teachers" will be used to represent this group). The inclusion criteria include teachers who participate in Thrive or Inspire Professional Learning in 2018-2019. Additionally, 449 teachers from 81 district schools (that are part of the Thrive and Inspire Professional Learning) are were randomized into the study will participate.
* To be eligible for the study, sites met the following criteria: a) have 2 or more PKFA classrooms; b) serve a high-need population and c) leaders ranked Thrive or Inspire as a first or second preference for the school. "High need" was defined as follows: the site level percentage of students in poverty was above the median of the eligible pool; the site level percentage of students in poverty was in the second quartile of the eligible pool and two or more students were listed as living in temporary housing; and/or the site level percentage of students in poverty was in the first quartile of the eligible pool and 5 or more students were listed as living in temporary housing.

Exclusion Criteria:

* Sites that were currently implementing ParentCorps at the time of the randomization were not eligible for the study. Only teachers who were part of the Thrive or Inspire Professional Learning tracks in 2018-2019 will be eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire-Modified (ERQ) | 1 Year
  Respondents indicate their tendency toward reappraisal (six items) and suppression (four items) through a seven-point Likert scale, ranging from one (strongly disagree) to seven (strongly agree). Independent scores are computed for each ER strategy. The ERQ had high internal consistency for both the cognitive reappraisal and expressive suppression subscales (α = .79 and .73, respectively) in a sample of undergrad students. The higher the scores the greater the use of the emotion regulation strategy.
Panorama Teacher and Staff Survey | 1 Year
  The survey exists as a series of scales, or sets of survey questions related to a single topic (e.g., Teaching Efficacy, Staff-Family Relationships or Educating all Students). The instrument was developed based on modern principles of survey design to substantially minimize measurement error. Some of these principles include wording items as questions, avoiding response options that may introduce acquiescence bias, avoiding double-barreled items, and using a variety of response options to capture a wider range of perceptions. This survey is currently in the process of being evaluated to accumulate evidence that the questions, scales, and instruments are reliable and valid.
Mindfulness in Teaching Scale-Modified | 1 Year
  used to assess the unique ways in which mindfulness may manifest in intrapersonal and interpersonal behaviors of teachers in a K-12 school setting. The original form of the self report measure is composed of two factors, "intrapersonal" and "interpersonal" mindfulness,and is a 14-item scale. The interpersonal sub scale has shown to predict teacher burnout (emotional exhaustion, de personalization) and instructional efficacy in working with students (social-emotional and behavioral management) over time. Cronbach Alpha internal consistency coefficients were found to be .861 for "Intrapersonal Mindfulness" and .711 for "Interpersonal Mindfulness." Higher score indicates more positive teaching behavior.
Parental Engagement of Families from Latino Backgrounds Questionnaire-Modified [PEFL- English] | 1 Year
  a 43-item Likert-type measure. The PEFL explores four dimensions of parental engagement related to children's school readiness: foundational education, supplemental education, school participation, and future-oriented teaching. The higher the average score on that scale, the more parents have agreed with the positive statements in the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Brotman, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States